CLINICAL TRIAL: NCT03985189
Title: A Japanese Phase 1 Study of ME-401 in Subjects With Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma and Roll Over Study for Subjects Who Have Participated in ME-401-004 Study
Brief Title: Study of ME-401 in Subjects With Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-401-K01
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory Indolent B-cell Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence | interventions — ME-401

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ME-401 (Experimental): ME-401 administered orally
  Interventions: Drug: ME-401

INTERVENTIONS:
Drug: ME-401 — [Phase 1 study (DLT evaluation)] ME-401 will be administered at 2 dosages as 45 mg (Cohort 1) or 60 mg (Cohort 2), daily oral administration, QD, and the trial will be initiated at Cohort 1, and medical specialists and the Efficacy and Safety Assessment Committee as needed will decide whether the Cohort will be shifted to the next stage based on their assessment of the safety and tolerability.
  [Roll over study] 60 mg ME-401 will be administrated on intermittent schedule (1 week on and 3 week off in every 4-week cycle)and will continue until the prescribed mediation in ME-401-004 study is completed or discontinuation criteria are met.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of ME-401 in the treatment of Japanese participants with Relapsed or Refractory indolent B-Cell Non-Hodgkin's Lymphoma and to continue administraion of ME-401 to patients with relapsed or refractory B-cell NHL with collecting safety information

ELIGIBILITY:
Inclusion Criteria:

[Phase 1 study (DLT evaluation)]

* Patients aged 20 years or older at the submission of the written informed consent form
* Patients with relapsed or refractory B-cell NHL
* Patients who have not undergone phosphatidylinositol 3-kinase inhibitor (PI3K) to date.
* Patients who have undergone Bruton's tyrosine kinase (BTK) inhibitors and have had no exacerbation during the use of BTK inhibitors.
* Patients with ECOG PS 0 or 1.

Exclusion Criteria:

[Phase 1 study (DLT evaluation)]

* Patients who underwent any major surgical treatment within 4 weeks prior to the initiation of the investigational product.
* Patients with poorly controlled diseases. The followings are the examples but the diseases will not be limited to those.
* Patients in whom any of HBV antigen/antibody, HCV antibody, HIV antibody or HTLV-1 antibody will be positive at screening test.
* Patients with active interstitial lung disease or a history thereof.
* Patients who have received the investigational products other than ME-401, systemic chemotherapy or radiotherapy within 4 weeks prior to the initiation of ME-401.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Up to approximately 1 year

SECONDARY OUTCOMES:
[Phase 1 study (DLT evaluation)] Plasma concentration level of ME-401 | Up to approximately 2 years
[Phase 1 study (DLT evaluation)] Maximum plasma drug concentration (Cmax) | Up to approximately 2 years
[Phase 1 study (DLT evaluation)] Area under the plasma drug concentration time curve (AUC) | Up to approximately 2 years
[Phase 1 study (DLT evaluation)] Terminal half-life (t1/2) | Up to approximately 2 years
[Phase 1 study (DLT evaluation)] Efficacy of ME-401 as assessed by the objective response rate (ORR) | Up to approximately 2 years
[Phase 1 study (DLT evaluation)] Efficacy of ME-401 will be assessed by the duration of response (DOR) | Up to approximately 2 years
[Phase 1 study (DLT evaluation)] Efficacy of ME-401 will be assessed by the progression-free survival (PFS) | Up to approximately 2 years
[Phase 1 study (DLT evaluation)] Efficacy of ME-401 will be assessed by the time to response (TTR) | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (9):
- Japan (9):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya, Aichi-ken
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tokyo Metropolitan Komagome Hospital, Bunkyo-ku, Tokyo
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
  - Aomori Prefectural Central Hospital, Aomori
  - Kyushu University Hospital, Fukuoka
  - Okayama University Hospital, Okayama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goto H, Izutsu K, Ennishi D, Mishima Y, Makita S, Kato K, Hanaya M, Hirano S, Narushima K, Teshima T, Nagai H, Ishizawa K. Zandelisib (ME-401) in Japanese patients with relapsed or refractory indolent non-Hodgkin's lymphoma: an open-label, multicenter, dose-escalation phase 1 study. Int J Hematol. 2022 Dec;116(6):911-921. doi: 10.1007/s12185-022-03450-5. Epub 2022 Sep 15. PMID 36107394
- See also: Goto H, Izutsu K, Ennishi D, et al. Zandelisib (ME-401) in Japanese patients with relapsed or refractory indolent non-Hodgkin's lymphoma: an open-label, multicenter, dose-escalation phase 1 study. Int J Hematol. 2022 Dec;116(6):911-921. — http://pubmed.ncbi.nlm.nih.gov/36107394/